CLINICAL TRIAL: NCT03918941
Title: Carey, a Mobile Coach Application for Patients Undergoing Orthognathic Surgery: a Multi-center Prospective Single Blind Randomized Clinical Trial About Patietn Information and Patient Satisfaction
Brief Title: Carey, a Mobile Coach Application for Patients Undergoing Orthognathic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Data Nurse, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Carey v 1.0
Record Dates: First submitted 2019-01-11; First posted 2019-04-18 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Dysgnathia
Keywords: patients satisfaction; Mobile application; orthognathic surgery

STUDY DESIGN:
Intervention Model Description: group 1 will use the mobile application (Carey) throughout their pre- and postoperative journey group 2 will follow the conventional pre- and postoperative care sequence (control group).
Who Masked: Investigator
Masking Description: The investigator does not know the identity of the patients neither which group uses the app
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carey (Experimental)
  Interventions: Device: Carey; Other: conventional information
- conventional information (Active Comparator)
  Interventions: Device: Carey; Other: conventional information

INTERVENTIONS:
Device: Carey — mobile application
Other: conventional information — leaflet, internet link and oral information

SUMMARY:
Carey is a mobile application guiding patients throughout their orthognathic surgery journey. The purpose of the application is optimizing the patient's experience before, during and after orthognathic surgery improving patient satisfaction and reducing complications. This will be evaluated based on the following outcomes:

1. Patient satisfaction based on a questionnaire
2. Objective parameters (complications, oral hygiene, amount of contacts with department, relapse,...)
3. Patient-reported outcomes (PROM)

The objective of the study is to evaluate whether the use of a mobile coach application in orthognathic surgery can improve patient satisfaction and reduce complications.

DETAILED DESCRIPTION:
Different studies pointed out the importance of patient information prior, during and after orthognathic surgery. It results in better recovery, less postoperative complications and improved patient satisfaction. In other words: a higher health care quality. Insufficient or omitted information about the procedure, surgical complications and/or postoperative care are an important cause of patient dissatisfaction.

Nowadays, patients receive a large amount of explanations, instructions and advices during their admission. Prior to surgery the surgeon will supply information about the procedure, sometimes aided by a website or online videos. Additionally the surgeon informs about the surgical complications, such as postoperative pain, restricted jaw movements, weight loss, swelling, scarring, jaw fixation, absenteeism from work, mood swings, and lip numbness.

The surgeon also supplies information by leaflets, oral and/or written instructions before discharge after surgery. This information however is often bulky, non-specific and incomplete. Furthermore, the surgeon knows that memory for medical information is poor and inaccurate resulting in nescient patients after returning home. For the surgeon it is a challenge to supply the right information at the right time, questioning the effectiveness of this conventional approach.

Some studies already showed that the use of multimedia represents a more effective method for patient education in comparison to the conventional approach. Patients prefer information through videos, interactive and moving images deriving better informed patients.

Furthermore, information provided by other patients was seen an added value. Adequate medication, dietary, oral hygiene and general advice could prevent complications.

Therefore, the use of interactive platforms such as a mobile application with phased information partition (the right information at the right time) could improve patient satisfaction, prevent unplanned consultations and even readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthognathic surgery
* Patients must be able to handle a smartphone.

Exclusion Criteria:

* Patients without smartphone
* Patients who have been submitted to orthognathic surgery in the past

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | At week 6
  Evaluation of patient satisfaction after surgery by means of a survey "Carey v1.0"

SECONDARY OUTCOMES:
Oral hygiene | At week 6 and 3 months postoperative
  By means of DPSI (Dutch periodontal screening index)
Pain control | At week 1 and week 3 postoperative
  By means of VAS (visual analogue scale: 0 no pain -10 pain)
Weight loss | the first 3 months postoperative
  Evaluation of patient weight in kilograms
Maximal mouth opening | At week 6 and 3 months postoperative
  Interincisal distance with a measuring rod in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Decoste, Drs, Principal Investigator — Universitair Ziekenhuis Brussel; Olivier Beckers, MD, Study Chair — Universitair Ziekenhuis Brussel; Maurice Mommaerts, Prof. Mult, Study Director — Universitair Ziekenhuis Brussel